CLINICAL TRIAL: NCT07078838
Title: A Randomized, Window of Opportunity Trial of Tirzepatide in Women With Obesity and a Diagnosis of Endometrial Intra-epithelial Neoplasia (EIN) or Grade 1 Endometrial Cancer
Brief Title: Tirzepatide in Women With Obesity and Endometrial Intra-epithelial Neoplasia or Grade 1 Endometrial Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2502; U01CA281026 (NIH)
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer; Endometrial Intraepithelial Neoplasia; Grade 1 Endometrial Endometrioid Carcinoma
Keywords: tirzepatide; obesity; tumor environment; cell proliferation
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia; Obesity; Hyperplasia | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- tirzepatide (Experimental): The treatment arm will receive 5mg tirzepatide for 4 weeks prior to standard of care surgery.
  Interventions: Drug: Tirzepatide
- No tirzepatide (No Intervention): No tirzepatide arm will not receive tirzepatide, and Standard Operating Procedures will be applied.

INTERVENTIONS:
Drug: Tirzepatide — Patients will receive a subcutaneous dose of 5 mg weekly for the 4 weeks prior to surgical staging.
  Arms: tirzepatide

SUMMARY:
The goal of this study is to determine the anti-proliferative effect of tirzepatide on the endometrium of patients with endometrial intra-epithelial neoplasia (EIN) and Grade 1 endometrial cancer (EC), by comparing archival endometrial biopsy samples of patients randomized to tirzepatide versus SOC (no tirzepatide) to their post-intervention hysterectomy specimens.

It was hypothesized that tirzepatide may help fight tumors in two ways: indirectly, by improving the body's overall metabolic health, and directly, by acting on abnormal cells in the uterus, such as those found in endometrial intraepithelial neoplasia (EIN) and endometrial cancer (EC). EIN is considered a precursor to EC. Tirzepatide may influence the tumor environment through key biological pathways related to insulin, fat metabolism, and mTOR signaling, all of which are often disrupted in individuals with obesity. Because both EIN and EC are strongly linked to obesity, tirzepatide could offer a promising dual benefit, promoting weight loss while also slowing or stopping tumor growth. The primary goal of this study is to determine whether tirzepatide can reduce cell proliferation in the lesions or tumors of patients with EIN and early- stage (Grade 1) EC.

Patients will either be randomized to receive tirzepatide or no tirzepatide for 4 weeks prior to their hysterectomy surgery. Patients randomized to the tirzepatide arm will be given a glucose monitoring system for continuous monitoring with real-time alarms to alert of hypoglycemia. Patients will complete diaries during treatment to document compliance with medication and record any side effects.

Patients will undergo standard of care surgery 7-10 days after the final dose of tirzepatide in order to minimize the risk of gastroparesis. During surgery (hysterectomy), an endometrial biopsy for uterine biopsy tissue will be collected.

At the 1-month post-operation visit, patients from both arms will be referred to an institutional weight loss clinic.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* The subject is willing and able to comply with study procedures based on the judgement of the investigator.
* Age > 18 years at the time of consent.
* ECOG ≤ 2 or Karnofsky Performance Status of >50
* Histological or cytological evidence/confirmation of endometrial intraepithelial neoplasia (EIN) or grade 1 endometrioid histology endometrial cancer (EC) and scheduled to undergo standard of care hysterectomy and staging.
* Subject must have archival EC tissue available.
* Body mass index of >30kg/m2
* Demonstrate adequate organ function as defined in the protocol, all screening labs to be obtained within 28 days prior to initiating study treatment

Exclusion Criteria:

* Active infection requires systemic therapy.
* Subject is pregnant or breast breastfeeding, or planning to become pregnant at any time during the study
* Taking any prescription medications or other drugs that influence weight change in the past 3 months.
* Known sensitivities (i.e., urticaria and eczema) to GIP and GLP-1 receptor agonists.
* Have type 1 diabetes mellitus or latent autoimmune diabetes in adults, or are receiving treatment with insulin.
* Have a history of severe hypoglycemia or not be able to communicate an understanding of hypoglycemic symptoms.
* Have a history of acute or chronic pancreatitis or serum lipase/amylase >2X ULN or fasting triglyceride >500 mg/dL at screening.
* Have a diagnosis of gastroparesis, history of bariatric surgery, or a clinically significant gastric emptying abnormality.
* Have a history or family history of multiple endocrine neoplasia, thyroid C-cell hyperplasia, or medullary thyroid carcinoma.
* Currently receiving another treatment for EIN or EC.
* Any condition, in the opinion of the investigator, which would prohibit safe participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Anti-proliferative effect of Tirzepatide | At 4th week (during surgery)
  Anti-proliferative effect of Tirzepatide will be measured via Immunohistochemistry analysis using multi-color fluorescence assays to assess Ki-67 staining.

SECONDARY OUTCOMES:
The Ki-67/caspase-3 ratio change | At 4th week (during surgery)
  The Ki-67/caspase-3 ratio will be assessed via immunohistochemistry, before and after treatment in the 2 groups. It is expected that the ratio will exhibit stronger intervention effects since proliferation should decrease and apoptosis should increase.
Response to treatment | At 4th week (during surgery)
  Response to treatment will be defined as a decrease of ≥13% in proliferation of the endometrium (EIN and EC) from pre- to post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Bae-Jump, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials